CLINICAL TRIAL: NCT05248906
Title: Giant Cell Arteritis - Examination of the Optimal Diagnostic Pathway
Brief Title: Giant Cell Arteritis - Optimization of Diagnostics
Acronym: GAME
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Steffen Hamann, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: H-20032069
Record Dates: First submitted 2020-11-03; First posted 2022-02-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2022-02

CONDITIONS: Giant Cell Arteritis
Keywords: Temporal artery biopsy,; Giant cell arteritis; Ultrasound; 18F-FDG PET/CT
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for DNA analysis will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Giant cell arteritis — Ultrasound 18F-fluorodeoxyglucose (18F-FDG) Positron Emission Tomography Temporal artery biopsy

SUMMARY:
Giant cell arteritis - Optimization of diagnostics

DETAILED DESCRIPTION:
A prospective study. Investigating the use of ultrasound, temporal artery biopsy, biomarkers and 18F-fluorodeoxyglucose positron emission tomography-computed tomography for establishing a diagnosis of giant cell (temporal) arteritis.

ELIGIBILITY:
Inclusion Criteria:

Clinical suspicion of giant cell arteritis

Meets the American College of Rheumatology Criteria:

Age at disease onset => 50 years New headache Temporal artery abnormality Elevated erythrocyte sedimentation rate >=50 mm/hour Abnomal artery biopsy

Exclusion Criteria:

Active cancer Use of steroid for more than a week (the prior 6 months)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical suspicion of giant cell arteritis
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Giant cell arteritis | Week 26
  Clinical verification of giant cell arteritis diagnosis as evaluated with a combination of ultrasound, biopsy and PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Hamann, MD, PhD,FEBO, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Klefter ON, Hansen MS, Lykkebirk L, Subhi Y, Brittain JM, Jensen MR, Dohn UM, Fana V, Wiencke AK, Heegaard S, Terslev L, Hamann S. Combining Paracentral Acute Middle Maculopathy and Peripapillary Fluid as Biomarkers in Anterior Ischemic Optic Neuropathy. Am J Ophthalmol. 2025 Mar;271:329-336. doi: 10.1016/j.ajo.2024.12.001. Epub 2024 Dec 6. PMID 39645178